CLINICAL TRIAL: NCT01522157
Title: A Randomized Cross-over Trial of the Postprandial Effects of Three Different Diets in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vårdcentralen Lyckorna (Other)
Responsible Party: Principal Investigator, Hans Guldbrand, Principal Investigator, Vårdcentralen Lyckorna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2011/418-31
Record Dates: First submitted 2012-01-17; First posted 2012-01-31 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diet; Low-carbohydrate; Postprandial; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Fat-Restricted; Diet, Carbohydrate-Restricted; Diet, Mediterranean

ARMS (1):
- All test patients (Active Comparator): All test patients are given low-fat, low-carbohydrate and mediterranean diet, in randomised order on different days.
  Interventions: Dietary Supplement: Low-fat Diet; Dietary Supplement: Low-carbohydrate Diet; Dietary Supplement: Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: Low-fat Diet — Low-fat Diet is provided for a breakfast and a lunch.
Dietary Supplement: Low-carbohydrate Diet — Low-carbohydrate Diet is provided for a breakfast and a lunch.
Dietary Supplement: Mediterranean Diet — Mediterranean Diet is provided for a breakfast and a lunch.

SUMMARY:
The trial will study the acute metabolic effects of three different types of diet: low-fat diet, low-carbohydrate diet and Mediterranean diet. About 20 patients with diabetes mellitus type 2 will be recruited and each of them will be given each type of diet on three different days. Menus with the same energy content but with different content of fat, carbohydrate and protein are designed. Breakfast and lunch are served for the patients each day of testing. Laboratory samplings are performed six times during the day. The order of the dietary intervention is randomized for each patient.

The investigators suppose to find different reaction in plasma glucose and lipids depending on the type of diet.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2

Exclusion Criteria:

* Treatment with insulin or sulfonylurea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
P-glucose | 6 months
  mmol/l
P-Triglycerides | 6 months
  mmol/l

SECONDARY OUTCOMES:
P-Cholesterol | 6 months
  mmol/l
P-LDL-Cholesterol | 6 months
  mmol/l
P-HDL-Cholesterol | 6 months
  mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nystrom, Professor, Principal Investigator — Department of Endocrinology Linköping University Hospital
Locations (1):
- Department of Medical and Health Sciences, Linköping University, Linköping, Sweden

REFERENCES:
- [Result] Fernemark H, Jaredsson C, Bunjaku B, Rosenqvist U, Nystrom FH, Guldbrand H. A randomized cross-over trial of the postprandial effects of three different diets in patients with type 2 diabetes. PLoS One. 2013 Nov 27;8(11):e79324. doi: 10.1371/journal.pone.0079324. eCollection 2013. PMID 24312178